CLINICAL TRIAL: NCT01564706
Title: Positron Emission Tomography Whole Body Biodistribution Using 18F-AV-45
Brief Title: A Study of 18F-AV-45 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Avid Radiopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18F-AV-45-A02
Record Dates: First submitted 2012-03-25; First posted 2012-03-28 (Estimated); Results first posted 2012-04-30 (Estimated); Last update posted 2012-05-18 (Estimated); Status verified 2012-05

CONDITIONS: Alzheimer Disease
Keywords: Amyloid imaging; Positron Emission Tomography; 18F-AV-45; florbetapir F 18; Diagnostic imaging
MeSH Terms: conditions — Alzheimer Disease | interventions — florbetapir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Healthy Volunteers (Experimental): Healthy male or female subjects, between 18 and 85 years of age.
  Interventions: Drug: florbetapir F 18

INTERVENTIONS:
Drug: florbetapir F 18 — IV injection, 370MBq (10mCi), single dose
  Other Names: 18F-AV-45; Amyvid; florbetapir

SUMMARY:
This study will determine how florbetapir F 18 (18F-AV-45) radioactivity is distributed throughout the body.

ELIGIBILITY:
Inclusion Criteria:

* Able to lie still on the imaging table for periods up to 1 hour

Exclusion Criteria:

* Radiation exposure for experimental purposes within the last year
* Claustrophobic or otherwise unable to tolerate the imaging procedure
* Medical condition or surgical history that would confound evaluation
* Current clinically significant cardiovascular disease
* Received an investigational medication within the last 30 days

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2007-10; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Avid Radiopharmaceuticals
Locations (1):
- Research Site, Jenkintown, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Volunteers: Single i.v. administration of approximately 10mCi 18F-AV-45
Period: Overall Study
Arm/Group | Healthy Volunteers
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 9
Age Continuous [Mean (Standard Deviation); unit: years] | 57.9 (10.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 3
Race/Ethnicity, Customized [Number; unit: participants]
  Black | 1
  Caucasian | 8
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Whole Body Radiation Dosimetry
Description: Radiation dose values (millisieverts/megabecquerel [mSv/MBq]) for regions of the whole body. Target organs included the adrenals, brain, breasts, gall bladder wall, lower large intestine wall, small intestine wall, stomach wall, upper large intestine wall, heart wall, kidneys, liver, lungs, muscle, ovaries, pancreas, osteogenic cells, skin, spleen, testes, thymus, thyroid, urinary bladder wall, uterus, and total body.
Time Frame: 0-380 min after injection
Measure: Mean (Standard Deviation); unit: mSv/MBq
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 9
mSv/MBq
  Effective Dose | 0.0186 (0.00426)
  Adrenals | 0.0136 (0.00129)
  Brain | 0.01 (0.00186)
  Breasts | 0.00624 (0.000865)
  Gallbladder Wall | 0.143 (0.0802)
  Lower Large Intestine Wall | 0.0278 (0.0102)
  Small Intestine | 0.0655 (0.0296)
  Stomach Wall | 0.0117 (0.000906)
  Upper Large Intestine Wall | 0.0745 (0.0342)
  Heart Wall | 0.0131 (0.00159)
  Kidneys | 0.013 (0.00111)
  Liver | 0.0644 (0.0221)
  Lungs | 0.00852 (0.000801)
  Muscle | 0.00863 (0.000762)
  Ovaries | 0.0176 (0.00434)
  Pancreas | 0.0144 (0.00134)
  Red Marrow | 0.0143 (0.00178)
  Osteogenic Cells | 0.0276 (0.00371)
  Skin | 0.00593 (0.000809)
  Spleen | 0.0089 (0.000986)
  Testes | 0.00681 (0.00129)
  Thymus | 0.00727 (0.00122)
  Thyroid | 0.00675 (0.00143)
  Urinary Bladder Wall | 0.0271 (0.0117)
  Uterus | 0.0156 (0.00319)
  Total Body | 0.0116 (0.000951)

ADVERSE EVENTS:
Time Frame: AEs occuring within 3 days of injection; SAEs occuring within 30 days of injection
Arm/Group | Healthy Volunteers
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 5/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Volunteers (N=9)
PALPITATIONS (Cardiac disorders) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 2 (2)
CHEST PAIN (General disorders) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 3 (3)
ANXIETY (Psychiatric disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days